CLINICAL TRIAL: NCT02281448
Title: Effect of BIA 2-093 on the Pharmacokinetics of a Combined Oral Contraceptive in Healthy Female Volunteers
Brief Title: Effect of BIA 2-093 on the Pharmacokinetics of a Combined Oral Contraceptive.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-114
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Results first posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate; Contraceptives, Oral, Combined

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment sequence A (Other): oral once daily dose of 1200 mg of BIA 2-093 plus single-dose of a contraceptive for 15 days followed by washout and 3 days of oral single-dose contraceptive
  Interventions: Drug: BIA 2-093; Drug: Contraceptives, Oral, Combined
- Treatment sequence B (Other): oral single-dose of a contraceptive for 3 days after pre-treatment with an oral once daily dose of 1200 mg of BIA 2-093 plus single-dose of a contraceptive for 15 days
  Interventions: Drug: BIA 2-093; Drug: Contraceptives, Oral, Combined

INTERVENTIONS:
Drug: BIA 2-093
Drug: Contraceptives, Oral, Combined

SUMMARY:
Single centre, two-way crossover, randomised, open-label study in 20 healthy female volunteers.The volunteers received an oral single-dose of a combined contraceptive containing with an oral once daily dose of 1200 mg of BIA 2-093

DETAILED DESCRIPTION:
Single centre, two-way crossover, randomised, open-label study in 20 healthy female volunteers.The volunteers received an oral single-dose of a combined contraceptive containing 30 μg ethinyloestradiol and 150 μg levonorgestrel on two occasions - once as such and once after pre-treatment with an oral once daily dose of 1200 mg of BIA 2-093 for 15 days separated by a washout period of at least 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal female;
* Able and willing to give written informed consent;
* Aged 18 to 40 years, inclusive;
* Not pregnant or breast-feeding;
* Body mass index (BMI) between 19 and 30 kg/m2, inclusive;
* Healthy as determined by medical history, physical examination, complete neurological examination, vital signs, and 12-lead ECG;
* Clinical laboratory tests with clinically acceptable results at screening and admission to the first period;
* Negative tests for HBsAg, anti-HCV Ab and HIV-1 and HIV-2 Ab at screening;
* Negative test for drugs of abuse at screening;
* Non-smoker or smokes less than 10 cigarettes or equivalent per day;
* Agreed to either practice abstinence or use a double-barrier or intra-uterine device from screening until the follow-up visit;
* Negative pregnancy test at screening and admission to the first period.

Exclusion Criteria:

* Had any contra-indication to the use of oral contraceptives;
* Had experienced notable adverse events while on any oral contraceptive;
* Had a history of alcoholism or drug abuse;
* Had a relevant history or presence of respiratory, gastrointestinal, renal, hepatic,haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders;
* Had acute gastrointestinal symptoms at the time of screening or admission to the first period;
* Had a significant infection or inflammatory process at the time of screening or admission to the first period;
* Had a relevant surgical history;
* Had a relevant family history;
* Had a history of relevant drug hypersensitivity (e.g., carbamazepine or oxcarbazepine);
* Had used relevant prescription or over-the-counter medication within 2 weeks ofadmission to the first period;
* Consumed more than 14 units of alcohol a week;
* Had participated in any clinical trial within 3 months prior to screening;
* Had previously received BIA 2-093;
* Had donated or received any blood or blood products within 2 months prior to screening;
* Was unlikely to co-operate with the requirements of the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-03; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- BIAL - Portela & Cª, S.A., S. Mamede Do Coronado, S. Mamede Do Coronado, Portugal

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence A: oral once daily dose of 1200 mg of BIA 2-093 plus single-dose of a contraceptive for 15 days followed by washout and 3 days of oral single-dose contraceptive
  BIA 2-093
  Contraceptives, Oral, Combined
- Treatment Sequence B: oral single-dose of a contraceptive for 3 days after pre-treatment with an oral once daily dose of 1200 mg of BIA 2-093 plus single-dose of a contraceptive for 15 days
  BIA 2-093
  Contraceptives, Oral, Combined
Period: Overall Study
Arm/Group | Treatment Sequence A | Treatment Sequence B
Started | 10 | 10
Completed | 8 | 9
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence A | Treatment Sequence B | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma BIA 2-194 Concentration
Description: Cmax - Maximum observed plasma BIA 2-194 concentration on days 1, 2, 4, 6, 8, 10, 12, 14 and 15 during a 15-day oral regimen of BIA 2-093 1200 mg once-daily.
Time Frame: Days 1, 2, 4, 6, 8, 10, 12, 14 and 15 during a 15-day oral regimen of BIA 2-093 1200 mg once-daily.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cmax (BIA 2-194): Mean trough (pre-dose) plasma concentrations of BIA 2-194 on Days 1, 2, 4, 6, 8, 10, 12, 14 and 15 during a 15-day oral regimen of BIA 2-093 1200 mg once-daily.
Arm/Group | Cmax (BIA 2-194)
Number analyzed (Participants) | 17
ng/mL
  Day 1 | 0.00 (0.00)
  Day 2 | 8443 (1422)
  Day 4 | 10691 (1736)
  Day 6 | 10961 (1737)
  Day 8 | 10175 (996)
  Day 10 | 10332 (1470)
  Day 12 | 10821 (1806)
  Day 14 | 10670 (1447)
  Day 15 | 9978 (1452)

2. Secondary Outcome: Cmax
Description: Cmax following administration of a single-dose of Microginon® concomitantly with the 14th dose of a 15-day oral regimen of BIA 2-093 1200 mg once-daily (Test) and following administration of a single-dose of Microginon® administered alone (Reference)
Time Frame: pre-dose, on Days 1, 2, 4, 6, 8, 10, 12, 14 and 15 of the BIA 2-093 + OC period.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Overall Population: Overall population - 17 subjects
Arm/Group | Overall Population
Number analyzed (Participants) | 17
pg/mL
  Cmax (ethinyloestradiol) Test | 53.4 (17.9)
  Cmax (ethinyloestradiol) Reference | 66.1 (19.1)
  Cmax (Levonorgestrel) Test | 3220 (1330)
  Cmax (Levonorgestrel) Reference | 3720 (1540)

3. Secondary Outcome: Tmax
Description: Tmax following administration of a single-dose of Microginon® concomitantly with the 14th dose of a 15-day oral regimen of BIA 2-093 1200 mg once-daily (Test) and following administration of a single-dose of Microginon® administered alone (Reference)
Time Frame: pre-dose, on Days 1, 2, 4, 6, 8, 10, 12, 14 and 15 of the BIA 2-093 + OC period.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Overall Population
Number analyzed (Participants) | 17
h
  tmax (ethinyloestradiol) Test | 1.67 (0.53)
  tmax (ethinyloestradiol) Reference | 1.52 (0.21)
  tmax (Levonorgestrel) Test | 1.28 (0.49)
  tmax (Levonorgestrel) Reference | 1.21 (0.36)

4. Secondary Outcome: AUC0-t
Description: AUC0-t (ng.h/mL) following administration of a single-dose of Microginon® concomitantly with the 14th dose of a 15-day oral regimen of BIA 2-093 1200 mg once-daily (Test) and following administration of a single-dose of Microginon® administered alone (Reference)
Time Frame: pre-dose, on Days 1, 2, 4, 6, 8, 10, 12, 14 and 15 of the BIA 2-093 + OC period.
Measure: Mean (Standard Deviation); unit: pg.h/mL
Arm/Group | Overall Population
Number analyzed (Participants) | 17
pg.h/mL
  AUC0-t (ethinyloestradiol) Test | 347 (145)
  AUC0-t (ethinyloestradiol) Reference | 595 (639)
  AUC0-t (Levonorgestrel) Test | 24000 (12100)
  AUC0-t (Levonorgestrel) Reference | 33600 (20000)

ADVERSE EVENTS:
Groups:
- Eslicarbazepine Acetate 1200 mg + Microginon®: Eslicarbazepine acetate 1200 mg + Microginon® (n=19)
- Microginon®: Microginon® (n=18)
Arm/Group | Eslicarbazepine Acetate 1200 mg + Microginon® | Microginon®
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 19/19 | 5/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eslicarbazepine Acetate 1200 mg + Microginon® (N=20) | Microginon® (N=20)
Abnormal values of neutrophils and white blood cells (Infections and infestations) | 1 (1) | 0 (0) — At discharge of her second treatment period (BIA 2-093 + Microginon®) 1 subject presented clinically relevant values for neutrophils and white blood cells count.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eslicarbazepine Acetate 1200 mg + Microginon® (N=19) | Microginon® (N=18)
Palpitations (Cardiac disorders) | 3 | 0
Eyelid oedema (Eye disorders) | 1 | 0
Abdominal colic (Gastrointestinal disorders) | 1 | 0
Change in bowel habits (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Epigastric fullness (Gastrointestinal disorders) | 1 | 0
Gastroenteritis noninfectious (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Xerostomia (Gastrointestinal disorders) | 1 | 0
Flu-like symptoms (General disorders) | 1 | 0
Increased thirst (General disorders) | 3 | 0
Thirst (General disorders) | 1 | 0
Escherichia coli cystitis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Catheter site ecchymosis (Injury, poisoning and procedural complications) | 3 | 0
Catheter site haematoma (Injury, poisoning and procedural complications) | 1 | 0
CPK increased (Investigations) | 1 | 0
Lymph node palpable (Investigations) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Concentration impairment (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 10 | 0
Facial paraesthesia (Nervous system disorders) | 1 | 0
Frontal headache (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 1
Incoordination (Nervous system disorders) | 1 | 0
Lightheadedness (Nervous system disorders) | 1 | 0
Paraesthesia lips (Nervous system disorders) | 3 | 0
Paraesthesia tongue (Nervous system disorders) | 1 | 0
Pre-syncope (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 14 | 0
Tremor of hands (Nervous system disorders) | 1 | 0
Vasovagal reaction (Nervous system disorders) | 2 | 1
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pain chest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acneiform eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema facial (Skin and subcutaneous tissue disorders) | 1 | 0
Erythematous eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Erythematous rash (Skin and subcutaneous tissue disorders) | 2 | 0
Generalized macular rash (Skin and subcutaneous tissue disorders) | 1 | 0
Localized erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes